Title: Treatment of Acute Pericarditis With Anakinra

NCT #: NCT03224585

Document approval date: June 8, 2017

Document Type: Statistical Analysis Plan

## STATISTICAL ANALYSIS PLAN

The primary endpoints will compare the change in pain score from baseline to 6 hours and baseline to 24 hours among all patients using a paired samples Wilcoxon test for nonparametric data.